CLINICAL TRIAL: NCT05440045
Title: A Phase 2, Multicenter, Open-Label Study to Evaluate the Preliminary Efficacy and Safety of 6MW3211 in Patients With Advanced Clear Cell Renal Cancer
Brief Title: A Clinical Study of 6MW3211 in Patients With Renal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6MW3211-2022-CP202
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-06

CONDITIONS: Advanced Clear Cell Renal Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 6MW3211 (Experimental): 6MW3211 injection, 30mg/kg
  Interventions: Drug: 6MW3211

INTERVENTIONS:
Drug: 6MW3211 — 6MW3211 injection, 30mg/kg, Q2W
  Other Names: 6MW3211 injection

SUMMARY:
single arm, non-randomized, multicenter, open label, phase 2 clinical trial in patients with advanced clear cell renal cacer

DETAILED DESCRIPTION:
This study is a single arm, non-randomized, multicenter, open label, phase 2 clinical trial to evaluate preliminary efficacy and safety in patients with advanced clear cell renal cacer

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the study and sign the informed consent.
* Advanced clear cell renal cancer.
* At least one measurable tumor target lesion.
* Life expectancy≥3 months.
* Suitable organ functions.
* Patients who had failed at least one line therapy.
* ECOG 0-1.
* The samples of tumor tissue should be provided

Exclusion Criteria:

* Patients who had received anti-tumor therapy/radiotherapy/immunotherapy within 4 weeks.
* History of other malignant tumors within 5 years.
* Patients with CNS metastasis.
* History of active autoimmune diseases.
* Patients with poor-controlled systemic diseases after treatment.
* Patients with severe infection or requiring antibiotic treatment within 4 weeks before dosing.
* Adverse reactions related to previous treatments failed to recover to CTCAE 5.0 ≤1
* Patients who had experienced immune-related adverse events (irAE) with grade 3 or above.
* Patients who were allergic to any composition of experimental drug.
* Subjects with poor treatment compliance.
* Pregnant or lactating woman.
* Live vaccination within 28 days before first dosing.
* History of drug abuse or addiction
* Patients with active HBV or HCV, or HIV antibody positive,or Tp-Ab positive.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 24 months
  Objective response rate